CLINICAL TRIAL: NCT07336485
Title: Impact of Forced Diuresis on the Residual Fragment Rate After Flexible Ureteroscopy for Management of Medium Sized Renal Stones
Brief Title: Forced Diuresis After Flexible Ureteroscopy for Medium-Sized Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Nasser Karamany Mokhat, Resident of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 685/2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stones
Keywords: Kidney stones; renal calculi; nephrolithiasis; flexible ureteroscopy; ureteroscopy; laser lithotripsy; residual stone fragments; stone-free rate; forced diuresis; furosemide; non-contrast computed tomography
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a one-to-one ratio to receive either intravenous furosemide-assisted forced diuresis during flexible ureteroscopy or standard care without furosemide during flexible ureteroscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furosemide-Assisted Forced Diuresis During Flexible Ureteroscopy (Experimental): During flexible ureteroscopy, participants received intravenous furosemide 40 milligrams total, divided into 20 milligrams administered 5 minutes after induction of anesthesia and 20 milligrams administered 30 minutes after the start of the procedure.
  Interventions: Drug: Furosemide
- Standard Care During Flexible Ureteroscopy Without Furosemide (Active Comparator): Participants underwent flexible ureteroscopy and received standard perioperative and postoperative care without receiving intravenous furosemide or any other diuretic medication.
  Interventions: Other: Standard Care After Flexible Ureteroscopy Without Furosemide

INTERVENTIONS:
Drug: Furosemide — Intravenous furosemide was administered as a total dose of 40 milligrams during the procedure, divided into 20 milligrams given 5 minutes after induction of anesthesia and 20 milligrams given 30 minutes after the start of the procedure.
  Arms: Furosemide-Assisted Forced Diuresis During Flexible Ureteroscopy
Other: Standard Care After Flexible Ureteroscopy Without Furosemide — Participants received standard perioperative and postoperative management after flexible ureteroscopy without administration of furosemide or any other diuretic medication.
  Arms: Standard Care During Flexible Ureteroscopy Without Furosemide

SUMMARY:
This randomized controlled clinical trial evaluated whether furosemide-assisted forced diuresis during flexible ureteroscopy reduced the residual fragment rate and improved the stone-free rate after flexible ureteroscopy for management of medium sized renal stones measuring up to 30 millimeters. Adult patients undergoing flexible ureteroscopy for renal stones were randomized into two parallel groups: an experimental group that received intravenous furosemide during the procedure and a control group that received standard perioperative and postoperative care without furosemide. Stone-free status and residual fragments were assessed using non-contrast computed tomography performed four weeks after the procedure, and residual fragments were classified by fragment size. Secondary outcomes included operative time, length of hospital stay, postoperative complications, total urine output in the first 24 hours, and the need for additional treatments for significant residual stones.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients who underwent flexible ureteroscopy for renal stones measuring 30 millimeters or less.

Exclusion Criteria:

* Patients with active urinary tract infection.
* Patients with a history of previous open renal surgery or renal trauma.
* Patients with contraindications to anesthesia, such as severe cardiac disease, uncontrolled diabetes mellitus, or severe coagulation disorder.
* Patients with severe renal impairment, defined as an estimated glomerular filtration rate less than 30 milliliters per minute per 1.73 square meters.
* Patients with a single kidney.
* Patients with contraindications to furosemide administration.
* Patients with congenital renal anomalies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Stone-free rate on non-contrast computed tomography | Four weeks after flexible ureteroscopy
  Stone-free status was assessed using non-contrast computed tomography performed four weeks after the procedure. Residual fragments were classified into four grades: Grade A (no stones), Grade B (0 to 2 millimeters), Grade C (2.1 to 4 millimeters), and Grade D (greater than 4 millimeters, clinically significant residual stones).

SECONDARY OUTCOMES:
Operative time | During procedure
  Operative time was calculated from insertion of the ureteroscope into the urethra until completion of ureteral stent placement.
Length of hospital stay | From end of procedure to hospital discharge (up to 7 days)
  Length of hospital stay was calculated from the day of surgery to the day of discharge.
Postoperative hematuria | From end of procedure through 4 weeks post-procedure
  Hematuria was recorded after the procedure.
Postoperative urinary tract infection | Within 7 days post-procedure
  Postoperative urinary tract infection was assessed within seven days after the procedure using fever with urinary symptoms and or a positive urine culture with significant bacteriuria.
Postoperative pain score | Recovery room (PACU), postoperative day 1, and at discharge (up to 7 days)
  Postoperative pain was assessed using a numerical rating scale (NRS) from 0 to 10, where 0 indicates no pain and 10 indicates worst imaginable pain (higher scores = worse pain). Pain was recorded in the recovery room (PACU), on postoperative day 1 (during admission), and at discharge.
Need for auxiliary treatment for clinically significant residual stones | Up to four weeks after flexible ureteroscopy
  The need for auxiliary treatment for clinically significant residual stones was recorded, including extracorporeal shock wave lithotripsy or repeat ureteroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals (Urology Department), Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlay the reported results were planned to be shared with other researchers. The shared data were planned to include baseline characteristics, stone characteristics, intraoperative details, stone-free outcome on non-contrast computed tomography at four weeks, and postoperative outcomes including complications, pain scores, urine output in the first 24 hours, and need for auxiliary treatment. A data dictionary was planned to be provided.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data were planned to become available after completion of the study and acceptance of the thesis or publication of the primary results, and were planned to remain available for five years.
Access Criteria: Access was planned to be provided to qualified researchers upon reasonable request, after review of a brief proposal and analysis plan, and after execution of a data use agreement. Data were planned to be shared in a secure electronic format with de-identification applied.